CLINICAL TRIAL: NCT05950009
Title: Relationship Between Major Depression and Periodontal Diseases: Analytical Cross-sectional Study
Brief Title: Relationship Between Major Depression and Periodontal Diseases
Acronym: LeakyBraInCS
Status: Recruiting | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Other Study IDs: URI 106-260623
Record Dates: First submitted 2023-07-03; First posted 2023-07-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder; Periodontitis
MeSH Terms: conditions — Depressive Disorder, Major; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases _major depression patients: subjects with moderate or severe major depression, without severe suicide ideation, as characterized by the Patient Health Questionnaire (PHQ)-9 index (values of 9 or greater) and by the Structured Clinical Interview for DSM-5 - (SCID) will be selected.
  Interventions: Other: No intervention (observational studies)
- Controls: subjects without mental health pathologies identified by SCID, who present an PHQ-9 index of 5 or below will be included as controls.
  Interventions: Other: No intervention (observational studies)

INTERVENTIONS:
Other: No intervention (observational studies) — No intervention (observational studies)

SUMMARY:
Background: There are epidemiological and preclinical studies in vivo that support the biological plausibility of the association between periodontal diseases and major depression (DM), through the hypothesis of a "leaky mouth" by periodontitis as a source of neuroinflammation. Therefore, this association should be studied in depth in carefully designed cross-sectional studies in humans to specifically assess this relationship.

Objectives: Primary: determine if periodontitis can be associated with the development of DM. Secondary: (1) to estimate the prevalence of periodontal diseases (gingivitis and periodontitis) in patients with and without DM; (2) to determine whether oral, periodontal, and fecal (bacterial, viral, and fungal) metagenomic microbiomes, inflammatory mediators, and intestinal barrier integrity are associated with periodontal and mental health variables.

Material and method:

A cross-sectional analytical study with two groups is designed:

* Control group (without DM): subjects without known mental health pathologies will be included, who present a PHQ-9 index of 5 or less. They will be recruited from the control group of a population-based study PsychoBioma TRIAD (C.P. PSQ-19-2 - C.I. 19/474-E). They will be matched by age, gender, and socioeconomic status.
* Group of cases (MD patients): subjects with moderate DM will be selected, characterized by HPQ9 index values of 9 or higher. They will be selected among those patients who attend the Mental Health consultations associated with the San Carlos Clinical Hospital.

The study will consist of three visits:

* Visit in Mental Health Consultations: in this visit the subject will be evaluated to determine if he meets the eligibility criteria. You will be informed of the purpose of the study and you will be invited to participate and sign the informed consent. After that, a structured clinical interview for the DSM-IV (SCID) will be conducted and the subject will fill in a series of specific scales on a study-specific electronic device [Beck Depression Inventory (BDI); UCLA Loneliness Scale, Center for Epidemiologic Studies Depression scale [CES-D]; Childhood Trauma Questionnaire short form (CTQ-SF); The World Health Organization Quality of Life questionnaire (WHOQOL); Hamilton scale (HAM-D17); Global Assessment of Functioning (GAF) Scale].
* Dental School Visit: Subject will receive a comprehensive periodontal examination. A subgingival microbiological sample, a saliva sample and a blood sample will also be taken. The patient will be given a specific vial to collect stool samples.
* At the participant's home: the stool samples will be deposited by the participants at home in the specific collection vial.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years.
* For the case group (MD patients), subjects with moderate or severe major depression, without severe suicide ideation, as characterized by the Patient Health Questionnaire (PHQ)-9 index (values of 9 or greater) and by the Structured Clinical Interview for DSM-5 - (SCID) will be selected.
* For the control group, subjects without mental health pathologies identified by SCID, who present an PHQ-9 index of 5 or below will be included as controls.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Diabetes mellitus.
* Chronic conditions: HIV infection, chronic intake of NSAIDs.
* Comorbidity with other mental disorders: eating disorders, borderline personality disorders, bipolar disorders, schizophrenia and related disorders, and/or any mental serious disease other than major depression.
* Severe suicide ideation.
* Patients who had received periodontal treatment for periodontitis in the last year.
* Presence of necrotizing periodontal diseases.
* Presence of less than three teeth per quadrant.
* Antibiotic use in the last 6 months prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects in the case group - MD group- will be selected from those patients seen at the Outpatient Clinic of Institute of Psychiatry and Mental Health of Hospital Clínico San Carlos.
  Subjects in the control group - Non MD group- will be recruited from the control group of a population-based study PsicoBioma TRIAD (C.P. PSQ-19-2 - C.I. 19/474-E) that is currently being performed by the lab of JCL. They will be matched on age, gender, and socio-economic status. In order to confirm that they are in good mental health, they will receive a pre-screen, online questionnaire to screen for symptoms of anxiety and depression (PHQ-9, STAI).
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Periodontitis (presence/absence) | Baseline
  With the clinical and radiological information, the periodontal diagnosis of the patients will be established according to the 2018 classification of periodontal and peri-implant diseases), which involves determining the stage (I to IV), the extent of the stage (localized, generalized or incisor-molar pattern) and the grade (A, B or C).

SECONDARY OUTCOMES:
Childhood Trauma Questionnaire short form (CTQ-SF) | Baseline
  Range: 25 to 125. A higher score means more (and worst) traumatic experience.
UCLA Loneliness Scale (Spanish version) | Baseline
  Range: 20 to 80. Higher scores indicatehigher levels of loneliness
The World Health Organization Quality of Life questionnaire (WHOQOL) | Baseline
  Range: 0 to100. A higher score means better quality of life.
Beck Depression Inventory (BDI) | Baseline
  Range: 0 to 63. A higher score means more severe-depressive symptomatology
Centre for Epidemiologic Studies Depression scale [CES-D] | Baseline
  Range: 0 to 60. Higher scores indicate the presence of more severe symptomatology
Hamilton scale (HAM-D17) | Baseline
  Range: 0 to 52. The higher the score, the more severe the depressive symptoms
Global Assessment of Functioning (GAF) Scale. | Baseline
  Range: 1 to 100. A higher score means better functioning. A score of 0 means Inadequate information.
Subgingival microbiota | Baseline
  Bacterial DNA extraction will be performed using a commercial kit (Molzym Gmbh& Co.KG; Bremen, Germany) specific for bacterial DNA extraction. DNA samples will be frozen at -80°C and preserved until further analysis by quantitative polymerase chain reaction (q-PCR) (Marin et al., 2019) and 16S rRNA sequencing, using the Illumina MiSeq platform. The analysis of sequences obtained for the microbiome will include: a) quality control and trimming: PCR primers, chimeric sequences, and short and low-quality reads will be discarded; b) mapping: annotation at different taxonomic levels; c) rarefaction curves; d) quantification: counts and percentages of the presence of specific bacteria in each sample at different taxonomic levels; e) calculation of the biodiversity index and f) comparison between samples. The analysis by q-PCR will include the detection and quantification of the most prevalent or abundant species.
Plasma levels of inflammatory mediators | Baseline
  plasma levels of inflammatory mediators IL-1β, TNF-α, IL-6, prostaglandin E2 and CPRhs
Saliva microbiota | Baseline
  microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences are compared to phylogenetic and functional databases to obtain taxonomic and functional profiles
Gut microbiota (Stool samples) | Baseline
  microbial DNA will be used for library preparation and metagenomic shotgun sequencing using the Illumina HiSeq 2500 System. Shotgun metagenomic sequencing can identify bacteria, fungi, and viruses, with a resolution that allows species-level identification. Sequences are compared to phylogenetic and functional databases to obtain taxonomic and functional profiles

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid
  - Instituto de Psiquiatría y Salud Mental, Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No